CLINICAL TRIAL: NCT03469388
Title: Arterial Stiffness, Blood Pressure and Cardiac Output Study; ABC-study A Prospective, Multidisciplinary Study of Arterial Stiffness Measures in Patients Treated for Aortic Aneurysms in Relation to Blood Pressure and Cardiac Output
Brief Title: Arterial Stiffness, Blood Pressure and Cardiac Output Study
Acronym: ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, MD, PhD, Rijnstate Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0820; NL57153.091.16 (Other: CMO-Arnhem Nijmegen)
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Infrarenal Abdominal Aortic Aneurysm
Keywords: EVAR, central pressure, arterial stiffness, AAA, elective surgery
MeSH Terms: interventions — Pulse Wave Analysis

STUDY DESIGN:
Intervention Model Description: prospective,multidisciplinary single center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elective EVAR patients (Experimental): Elective EVAR patients will be included in one arm only
  Interventions: Diagnostic Test: Pulse wave analyses; central blood presaure parameters

INTERVENTIONS:
Diagnostic Test: Pulse wave analyses; central blood presaure parameters — Pulse wave analyses; central blood presaure parameters
  Other Names: Pulse wave velocity

SUMMARY:
Comparison of non-invasively obtained central blood pressure using SphygmoCor and invasively recorded central blood pressure in patients with an AAA that will be treated with EVAR.

DETAILED DESCRIPTION:
Primary objective of the first study: validation of non-invasive central pressure parameters in patients treated with EVAR against invasive measurements.

Objectives of subsequent studies: Do non-invasive central parameters change over time after EVAR? What is the influence of intraluminal thrombus (presence, amount, configuration) on non-invasive central pressure parameters (and other obtained parameters of arterial stiffness)? Prospective study with consecutive, eligible subject enrollment. All subjects will undergo the Endovascular Aneurysm repair procedure with an endovascular device. Subjects will be followed procedurally, at 6-8 weeks and 1 year post implantation.

This study is a collaboration of the following departments of the Vascular Center in the Rijnstate Hospital Arnhem: Vascular Surgery, Interventional radiology, Internal Vascular Medicine, Cardiology.

Patients diagnosed with an abdominal aortic or aortoiliac aneurysm who are considered candidates for endovascular repair and who meet the study eligibility criteria may be screened for enrollment in the study. Up to 20 subjects will be enrolled .

Pre-procedural high resolution, contrast-enhanced CT scan evaluation to determine anatomical eligibility for enrollment will be performed within three months of the study procedure, according to standard care. Following EC/IRB approval of the study and the written informed consent form, patients will be screened for eligibility. Following informed consent, clinical characteristics will be reported (from hospital records). Per-procedural PWA measurements will be performed simultaneously with intravascular pressure measurements pre-implantation and after completion of the endocasular implantation. Subjects will be followed at 30 days and 1 year post-implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old;
2. Informed consent form understood and signed and patient agrees to follow-up visits;
3. Have a infrarenal abdominal aortic aneurysm (AAA) with maximum sac diameter ≥ 5.5cm, or an AAA ≥ 4.5 cm which has increased by > 1.0 cm in the past year with a scheduled endovascular intervention

Exclusion Criteria:

1. Life expectancy < 2 years;
2. Psychiatric or other condition that may interfere with the study;
3. Participating in another clinical study, interfering on outcomes;
4. Irregular pulse;
5. Presence of extensive peripheral arterial disease (ABI < 0.9 or obstruction validated on imaging); dated less than 3 months prior to treatment
6. Ruptured, leaking or mycotic aneurysm;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
central blood pressure | one week
  comparison of invasively recorded and non-invsively estimated central blood pressure

SECONDARY OUTCOMES:
changes in arterial stiffness pre- and post EVAR | 1 year
  changes in arterial stiffness pre- and post EVAR
influence of thrombus on arterial stiffness | 1 year
  influence of thrombus on arterial stiffness
changes in arterial stiffness over time | 1 year
  changes in arterial stiffness over time

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, PhD, Principal Investigator — Rijnstate
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Holewijn S, Vermeulen JJM, van Helvert M, van de Velde L, Reijnen MMPJ. Validation of Central Pressure Estimation in Patients with an Aortic Aneurysm Before and After Endovascular Repair. Cardiovasc Eng Technol. 2022 Apr;13(2):265-278. doi: 10.1007/s13239-021-00574-3. Epub 2021 Sep 28. PMID 34585343